CLINICAL TRIAL: NCT03240562
Title: Ultrasound-guided Serratus Anterior Plane Block for Thoracic Surgery Pain?
Brief Title: Ultrasound-guided Block for Thoracic Surgery Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMC2017-06-123
Record Dates: First submitted 2017-07-28; First posted 2017-08-07 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Pain; Thoracic Cancer
Keywords: serratus anterior plane block; ultrasound-guided; regional anesthesia; thoracic surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV-PCA group (Sham Comparator): no block performing, only use intravenous patient controled analgesia(IV-PCA)
  Interventions: Drug: patient controlled analgesia
- SAPB group (Experimental): serratus anterior plane block(SAPB) and intravenous patient controled analgesia(IV-PCA)
  Interventions: Procedure: serratus anterior plane block; Drug: patient controlled analgesia

INTERVENTIONS:
Procedure: serratus anterior plane block — before surgery :ultrasound-guided serratus anterior plane block
  Arms: SAPB group
Drug: patient controlled analgesia — two groups have same intravenous patient controlled analgesia

SUMMARY:
The investigators aimed to assess Ultrasounde- guided serratus anterior plane block can be effective in acute postoperative pain following thoracic surgery.

DETAILED DESCRIPTION:
Analgesic options for thoracotomy are various with each having their own merits and demerits.Thoracic epidural is said to be the gold standard for management of thoracotomy pain. However, it is invasive procedure and many side effects. Other options include paravertebral block, interpleural block, intrathecal opioids. Especially, paravertebral block is thought good alternative to epidural anethesia. Most of these invasive neuraxial techniques demand normal coagulation parameters to be present.

The serratus anterior plane block(SAPB) was done under ultrasound guidance in the mid-axillary line at the level of the fourth rib and the catheter was placed superficial to the serratus plane. The patient expressed relief in pain within 10 minutes of being given the bolus of local anaesthetic.Pain following thoracotomy is chiefly due to rib retraction, and damage to the serratus/intercostal muscles and intercostal nerves. A SAPB addresses both these aspects. SAPB has been mentioned in previous studies for management of rib fractures and breast surgeries. The investigators try to evaluate whether the SAPB is easy to perform and provides effective analgesia in patients undergoing thoracotomy with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

•undergoing thoracic surgery (lobectomy or segmentectomy)

Exclusion Criteria:

• allergy to any drugs chronic pain disease with medication psychologic disorder anti-depressant drug chronic kidney disease ( Cr over 2.0 mg/dl) coagulopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
opioid consumption | the first 24hour in postoperative phase
  the dose of PCA and residual opioid

SECONDARY OUTCOMES:
postoperative pain scale | intraoperative(immediately after surgery), postoperative 6 ,12, 24 hour
  numeric rating scale
opioid consumption | the first 6,12 hour in postoperative phase
  the dose of PCA and residual opioid

OTHER OUTCOMES:
questionnaire about patient's satisfaction for pain management | postoperative 24 hour
  score 1(bad)-5(good)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu GM, Jarvis GC. Serratus Anterior Plane Block to Address Postthoracotomy and Chest Tube-Related Pain: A Report on 3 Cases. A A Case Rep. 2017 Jun 15;8(12):322-325. doi: 10.1213/XAA.0000000000000502. PMID 28614112
- [Background] Duceau B, Baubillier M, Bouroche G, Albi-Feldzer A, Jayr C. Pupillary Reflex for Evaluation of Thoracic Paravertebral Block: A Prospective Observational Feasibility Study. Anesth Analg. 2017 Oct;125(4):1342-1347. doi: 10.1213/ANE.0000000000002003. PMID 28489642
- [Background] Liu F, Zhang H, Zuo Y. Bilateral thoracic Paravertebral block for immediate postoperative pain relief in the PACU: a prospective, observational study. BMC Anesthesiol. 2017 Jul 5;17(1):89. doi: 10.1186/s12871-017-0378-3. PMID 28679359
- [Background] Terkawi AS, Tsang S, Sessler DI, Terkawi RS, Nunemaker MS, Durieux ME, Shilling A. Improving Analgesic Efficacy and Safety of Thoracic Paravertebral Block for Breast Surgery: A Mixed-Effects Meta-Analysis. Pain Physician. 2015 Sep-Oct;18(5):E757-80. PMID 26431130
- [Background] Wildgaard K, Petersen RH, Hansen HJ, Moller-Sorensen H, Ringsted TK, Kehlet H. Multimodal analgesic treatment in video-assisted thoracic surgery lobectomy using an intraoperative intercostal catheter. Eur J Cardiothorac Surg. 2012 May;41(5):1072-7. doi: 10.1093/ejcts/ezr151. Epub 2011 Dec 21. PMID 22219442
- [Background] Madabushi R, Tewari S, Gautam SK, Agarwal A, Agarwal A. Serratus anterior plane block: a new analgesic technique for post-thoracotomy pain. Pain Physician. 2015 May-Jun;18(3):E421-4. PMID 26000690